CLINICAL TRIAL: NCT01712386
Title: The Effects of Dietary Nitrate Supplementation on the Oxygen Cost of Moderate-Intensity Exercise and Functional Capacity in Mild-Moderate COPD Patients
Brief Title: Nitrate, Chronic Obstructive Pulmonary Disease (COPD) and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIHR Exeter Clinical Research Facility (Network)
Collaborators: Torbay and South Devon NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 12/SW/0327; PC/jse (Other Grant/Funding Number: Torbay Medical Research Fund)
Record Dates: First submitted 2012-10-12; First posted 2012-10-23 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- COPD (Experimental)
  Interventions: Dietary Supplement: Beetroot; Dietary Supplement: Beetroot placebo

INTERVENTIONS:
Dietary Supplement: Beetroot
  Other Names: James Whites Drinks beetroot sports shot
Dietary Supplement: Beetroot placebo
  Other Names: James Whites Drinks beetroot sports shot

SUMMARY:
Patients with moderate chronic obstructive pulmonary disease (COPD) typically have reduced exercise capacity. This is because their lungs are damaged and because of increased work of breathing. In some patients, exercise capacity is reduced to such a level that even simple activities of daily living, such as washing and dressing, may impose a challenge.

Recent findings in healthy young people suggest that increasing the amount of nitrate in our diet in the form of beetroot juice can improve the ability to exercise. Studies involving cycling have shown that less oxygen is needed to perform the same level of exercise after taking more nitrate in the diet. Nitrate (found in abundance in beetroot) is known to be converted in the body to nitric oxide (NO), a substance which increases blood flow and may affect the energy-producing mechanisms inside muscle cells. A recent exciting finding is that such dietary nitrate supplementation appears to reduce the amount of oxygen needed to complete moderate intensity exercise (walking) in healthy individuals. It is the purpose of this study to see if such effects could be seen in COPD patients. If this is indeed the case, then it may suggest that a period of dietary supplementation of a relatively cheap, widely available, and natural food product may improve the ability of patients to undergo everyday tasks and ultimately improve their quality of life.

To help investigators understand the effects of dietary nitrate supplementation on the ability to exercise in COPD patients, the investigators will recruit 15 people with mild to moderate disease. They will complete a series of undemanding exercise tests on three separate occasions. On one occasion they will have had a course of nitrate rich beetroot juice leading up to the tests, and on the other occasion they will have had a course of beetroot juice with the nitrate removed. The investigators will monitor blood pressure, levels of nitrate and nitrite in the blood, oxygen uptake and functional capacity during the tests which will allow us to assess any effects that may have occurred as a result of increased nitrate intake.

ELIGIBILITY:
Inclusion Criteria:

* Mild-moderate COPD (FEV1 30%-80% predicted values)
* Between the ages of 40-75
* Able to give informed consent

Exclusion Criteria:

* Uncontrolled hypertension (systolic BP> 160mmHg, diastolic >100mmHg)
* Regular therapy with organic nitrates, nicorandil and antibiotics.
* Current smoker (Have smoked within the last 3 months)
* Chronic Kidney Disease (stage 4 or worse)
* Any other serious medical condition which would interfere with data interpretation and safety or that may make cycling exercise difficult, limited or uncomfortable.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
O2 cost of moderate-intensity cycling exercise | Twice over a maximum of a 2 month period
  whether nitrate reduces the O2 cost of moderate intensity exercise.

SECONDARY OUTCOMES:
Single-breath lung diffusion capacity | Once at screening. i.e. on one day that will last 10 seconds (before should only have been at familiarisation)

OTHER OUTCOMES:
Functional capacity measured by 6-Minute Walking Test (6MWT) | Twice over a maximum of a 2 month period

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Benjamin, Professor, Principal Investigator — Torbay and South Devon NHS Foundation Trust
Locations (1):
- South Devon Healthcare NHS Foundation Trust, Torquay, Devon, United Kingdom